CLINICAL TRIAL: NCT02955732
Title: Bioavailability and Pharmacokinetics of Intranasal Dexmedetomidine in Children
Brief Title: Pharmacological Characteristics of Intranasally Given Dexmedetomidine in Paediatric Patients
Acronym: PINDEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T280/2016
Record Dates: First submitted 2016-11-03; First posted 2016-11-04 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Procedural Sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intranasal dex (Experimental): Dexmedetomidine 2-4 µg/kg alone
  Interventions: Device: Dexmedetomidine

INTERVENTIONS:
Device: Dexmedetomidine — A 2-4 µg/kg dose of the study drug, 2 µg/kg of intranasal dexmedetomidine, will be administered using a LMA MAD Nasal™ -device approximately 20 min prior to planned sedation/anesthesia.
  Other Names: Dexdor

SUMMARY:
We aim to characterize the bioavailability and pharmacokinetics of dexmedetomidine after intranasal dosing employing pharmacometrics methods in otherwise healthy 1 month to 11 years of age children scheduled for minor surgery or other procedures requiring sedation or anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 1. The child is scheduled for intra-articular drug injections, hernia repair, bronchoscopy or another similar minor procedure or magnetic resonance imaging requiring sedation or anesthesia
* 2. Guardians and patient (if relevant) with fluent skills in the Finnish or Swedish language (to understand the given information, to be able to give informed consent and communicate with the study personnel).
* 3. Age between 1 month and 12 years.
* 4. Normal developmental status including growth (SD -1.5-1.5)
* 5. Written informed consent from the guardian and the patient (when relevant).

Exclusion Criteria:

* 1. A previous history of intolerance to the study drug or to related compounds and additives
* 2. Prior drug therapy with dexmedetomidine in the 14 days prior to the study.
* 3. Use of any drugs known to cause enzyme induction or inhibition for a period of 30 days prior to the study, use of any natural products (including grapefruit products) for at least 14 days prior to the study and caffeine containing products for at least 24 hours prior to the study. The use of regular doses of paracetamol is allowed.
* 4. Existing or recent significant disease that could influence the study outcome or cause a health hazard for the subject if he/she would participate in the study.
* 5. Participation in any other clinical study involving investigational or marketed drug products concomitantly or within one month prior to the entry into this study.
* 6. Clinically significant abnormal findings in physical examination or laboratory screening [routine haematology (haemoglobin, haematocrit, red blood cell count, white blood cell count, platelets), renal function tests (creatinine, urea) and liver function tests (bilirubin)].

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-01-01; Primary Completion 2017-04-30 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability (%) of intranasally given dexmedetomidine | 4 hours

SECONDARY OUTCOMES:
Change in hemodynamic parameter (blood pressure) | 6 hours
  More than 30% change from the baseline in the blood pressure (measured in mmHg)
Change in hemodynamic parameter (heart rate) | 6 hours
  More than 30% change from the baseline in the heart rate (measured in beats per minute)
Number of patients with adverse events as a measure of safety and tolerability | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Panu Uusalo, MD, Principal Investigator — Dept. Anaesthesilogy and Intensive Care, University of Turku and Turku University Hospital
Locations (1):
- Perioperative Services, Intensive Care and Pain Therapy, Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No